CLINICAL TRIAL: NCT02028026
Title: The Effects of Vilazodone on Glutamate in the Anterior Cingulate Cortex in Anxious Unipolar Depressives
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit eligible subjects
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Michael Henry, Medical Director, Bipolar Clinic, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VII-IT-10; 2013P000335 (Other: Partners Human Research Office)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder; Anxiety; Comorbidity
Keywords: Depressive Disorder; Anxiety; Comorbidity; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Citalopram; Vilazodone; Serotonin Uptake Inhibitors; Receptor, Serotonin, 5-HT1A
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Depressive Disorder | interventions — Vilazodone Hydrochloride; Citalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vilazodone (Experimental): 10mg/day for 1 week, 20 mg/day for 1 week, and then 40 mg/day for 6 weeks.
  Interventions: Drug: Vilazodone
- Citalopram (Active Comparator): 20 mg/day for 2 weeks and then 40 mg/day for 6 weeks.
  Interventions: Drug: Citalopram

INTERVENTIONS:
Drug: Vilazodone — 10mg/day for 1 week, 20 mg/day for 1 week, and then 40 mg/day for 6 weeks.
  Other Names: Viibryd
  Arms: Vilazodone
Drug: Citalopram — 20 mg/day for 2 weeks and then 40 mg/day for 6 weeks
  Other Names: Celexa, Cipramil
  Arms: Citalopram

SUMMARY:
The purpose of this study is to determine whether vilazodone is more effective than citalopram for the treatment of anxious depression. We will use neuroimaging to see whether there are changes in the brains of patients receiving the drug vilazodone that are different from those of citalopram. These changes may show that vilazodone affects the brain differently than most other kinds of standard antidepressant medications.

DETAILED DESCRIPTION:
This study proposes to utilize recent advances in magnetic resonance spectroscopy (MRS) techniques that permit reliable measurement of Glu in humans (9) to examine whether Vilazodone and citalopram exert differential effects on Glutamatergic neurotransmission in the ACC of anxious unipolar depressed patients. Functional connectivity as measured by Blood Oxygen Level Dependent (BOLD) MRI will be assessed to determine the relationship between the change in connectivity and the change in Glu levels with treatment. We also propose to examine, in an exploratory fashion, the relative effect of the two drugs on BOLD activation in the insula cortex.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-50 years.
* Meets DSM-IV criteria for unipolar major depression.
* MADRS score > 20.
* Subject exhibits clinically significant anxiety and HAM-A score > 15.
* Capable of providing informed consent.
* Has an established residence and phone.

Exclusion Criteria:

* A clinically significant medical condition which could impact the response of the individual to antidepressant treatment (e.g. diabetes, cancer, lupus or other autoimmune illness). Stably treated hypothyroidism (TSH < 2) will be permitted.
* Beta blockers, antidepressants, antipsychotics, lithium, antiepileptic medications, steroids (oral and inhaled), chronic use of nonsteroidal antinflamatory medications (infrequent sporadic use permitted), or other medications with the potential to interfere with the antidepressant effects of Vilazodone.
* Pregnancy.
* In women of childbearing potential an unwillingness to use reliable methods to prevent pregnancy.
* History of manic or psychotic symptoms.
* History of seizure or epilepsy.
* History of alcohol or drug dependence and active use of substances in the past month.
* Active alcohol or drug abuse.
* Ingestion of 4 or more caffeinated beverages a day, on average.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Glutamate Levels | Week 0 and Week 4
  Our hypothesis that Vilazodone will increase ACC glutamate levels more than Citalopram will be addressed using a repeated measures linear regression model with ACC glutamate level as the outcome and drug (Vilazodone or Citalopram) and drug x scan time (baseline or follow-up) interaction as predictors.

SECONDARY OUTCOMES:
Functional Connectivity | Week 0 and Week 4
  Our hypothesis that Vilazodone will decrease functional connectivity more than Citalopram will be addressed using a repeated measures linear regression model with functional connectivity correlation as the outcome and drug (Vilazodone or Citalopram) and drug x scan time (baseline or follow-up) interaction as predictors.

OTHER OUTCOMES:
Change in BOLD signal | Week 0 and Week 4
  Exploratory analyses will estimate the effect size of the different treatments on change in BOLD signal.
Change in MADRS Score | Screen and Weeks 0, 2, 4, 6, & 8
  Associations with change in MADRS score will be quantified by incorporating treatment, change in glutamate level, change in functional connectivity, and their interactions with follow-up time as predictors in repeated measures linear regression models with MADRS scores as repeated outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Henry, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States